CLINICAL TRIAL: NCT00106587
Title: Treatment of In-Stent Restenosis by Paclitaxel Coated PTCA Balloons
Brief Title: Treatment of In-Stent Restenosis by Paclitaxel Coated PTCA Balloons (PACCOCATH - ISR I)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMT - Pac 1
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Coronary Restenosis
Keywords: in stent restenosis; paclitaxel coated balloon catheter; paccocath; drug eluting balloon
MeSH Terms: conditions — Coronary Restenosis | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Uncoated Angioplasty (Active Comparator): PTCA of ISR
  Interventions: Device: PTCA
- DCB Angioplasty (Experimental): DCB PTCA of ISR
  Interventions: Combination Product: paclitaxel coated balloon catheter (device with drug)

INTERVENTIONS:
Device: PTCA
  Arms: Uncoated Angioplasty
Combination Product: paclitaxel coated balloon catheter (device with drug)
  Arms: DCB Angioplasty

SUMMARY:
The PACCOCATH ISR study is a randomized, double-blinded German multicenter trial on the efficacy and tolerance of a paclitaxel coated balloon catheter in coronary in-stent restenosis.

DETAILED DESCRIPTION:
Background: Drug-eluting stents have shown promising anti-restenotic effects in clinical trials. It may be preferable, however, to avoid the stent-in-stent approach in treating in-stent restenosis (ISR). In prior animal trials, we demonstrated a highly significant reduction of neointimal formation by drug-eluting balloon catheters (DEB). The aim of the PACCOCATH ISR study is to investigate the novel DEB in the treatment of ISR.

Methods and results: The PACCOCATH ISR study is a randomized, double-blind German multicenter trial on the efficacy and tolerance of the DEB in coronary ISR. Patients are randomized to rePTCA of ISR either using the coated PTCA balloon (3 µg paclitaxel/mm² balloon surface) or a non-coated balloon of the same type (n=52 patients). Balloon inflation time is 60 seconds in both cases. Major inclusion criteria are an ISR in a coronary artery with a diameter stenosis of at least 70%, < 25 mm length, and a vessel diameter of 2.5 to 3.5 mm. The primary endpoint is late lumen loss after 6 months (independent angiographic core lab). Secondary endpoints are binary restenosis rate and major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical evidence of stable or unstable angina or a positive functional study
* Single, restenotic lesion in a stented coronary artery (allowed are multiple lesions but only the target lesion is amenable for percutaneous intervention, i.e. no 'staged' procedures involving non-target lesions)
* Diameter stenosis > 70% (visual estimate)
* Stented segment length < 25 mm
* Vessel diameter => 2.5 mm
* Female patients can enter this study if they are post-menopausal for at least two years or have undergone hysterectomy or sterilization
* Signed patient informed consent form
* Patients and treating physicians agree that the patient will return for all required post procedure follow-up assessments as defined in the clinical protocol

Exclusion Criteria:

* Left ventricular ejection fraction of < 30%
* Target lesion/vessel with any of the following characteristics: Clear angiographic calcification in the target lesion or greater than mild calcification in the proximal vessel (minimally radiopaque densities that are discrete and non-linear). Visible thrombus proximal to the lesion.
* Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, abciximab, paclitaxel, or a sensitivity to contrast media which cannot be adequately pre-medicated.
* Other medical illness (i.e. cancer, liver disease or congestive heart failure) that may require cytostatic or radiation therapy causing the subject to be non-compliant with the protocol, confound the data interpretation or is associated with limited life-expectancy (i.e., less than two years).
* Severe chronic renal insufficiency.
* Significant gastrointestinal (GI) bleed within the past six months. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Extensive peripheral vascular disease that precludes safe 6 French sheath insertion and/or requires additional anti-platelet and/or anti-coagulation treatment.
* Participating in another device or drug study within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
angiographic late lumen loss | 6 months
  angiographic late lumen loss

SECONDARY OUTCOMES:
binary restenosis rate | 6 months
  binary restenosis rate
major adverse cardiac events | 12 months
  major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, MD, Principal Investigator — Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, 66421 Homburg/Saar, Germany; Ulrich Speck, PhD, Study Director — Radiologie, Campus Mitte, Charite, Berlin, Germany
Locations (5):
- Germany (5):
  - Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, Homburg / Saar, Saarland
  - Kardiologie, Campus Mitte, Charite, Berlin
  - Kardiologie, Campus Virchow-Klinikum, Charite, Berlin
  - Medizinische Universitätsklinik III, Abt. Kardiologie und Angiologie, Freiburg im Breisgau
  - I. Medizinische Klinik, Universitaetsklinikum, Mannheim

REFERENCES:
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Speck U, Scheller B, Abramjuk C, Grossmann S, Mahnkopf D, Simon O. Inhibition of restenosis in stented porcine coronary arteries: uptake of Paclitaxel from angiographic contrast media. Invest Radiol. 2004 Mar;39(3):182-6. doi: 10.1097/01.rli.0000116125.96544.64. PMID 15076010
- [Background] Scheller B, Speck U, Schmitt A, Bohm M, Nickenig G. Addition of paclitaxel to contrast media prevents restenosis after coronary stent implantation. J Am Coll Cardiol. 2003 Oct 15;42(8):1415-20. doi: 10.1016/s0735-1097(03)01056-8. PMID 14563585
- [Background] Scheller B, Speck U, Romeike B, Schmitt A, Sovak M, Bohm M, Stoll HP. Contrast media as carriers for local drug delivery. Successful inhibition of neointimal proliferation in the porcine coronary stent model. Eur Heart J. 2003 Aug;24(15):1462-7. doi: 10.1016/s0195-668x(03)00317-8. PMID 12909076
- [Derived] Scheller B, Clever YP, Kelsch B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Speck U, Bohm M, Cremers B. Long-term follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. JACC Cardiovasc Interv. 2012 Mar;5(3):323-30. doi: 10.1016/j.jcin.2012.01.008. PMID 22440499
- [Derived] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Two year follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2008 Oct;97(10):773-81. doi: 10.1007/s00392-008-0682-5. Epub 2008 Jun 5. PMID 18536865
- [Derived] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615